CLINICAL TRIAL: NCT00134134
Title: An Open-Label Assessment of the Efficacy & Safety of Efalizumab in the Treatment of Moderate-Severe Hydradenitis Suppurativa
Brief Title: Efficacy and Safety of Efalizumab in the Treatment of Moderate-Severe Hydradenitis Suppurativa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H12452-01B
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Hidradenitis Suppurativa
Keywords: hidradenitis suppurativa; efalizumab; biologic; Raptiva
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — efalizumab

INTERVENTIONS:
Drug: efalizumab

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of efalizumab in treating hydradenitis suppurativa, and to evaluate the duration of the benefit seen in people who respond to treatment with efalizumab, after the medication is stopped.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the efficacy of subcutaneously administered efalizumab in the treatment of refractory, severe hydradenitis suppurativa. The secondary objectives of this study are to assess the ability to re-establish disease control after discontinuation of drug and allowance for relapse of disease, as well as to assess the safety of subcutaneously administered efalizumab in the treatment of refractory, severe hydradenitis suppurativa.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18-65 years of age
* Has Hydradenitis Suppurativa (HS) involving at least 1 area of the body with greater than or equal to 12 lesions; onset of disease is 6 months and greater.
* Failed at least 3 months of standard conventional therapies such as antibiotics and/or systemic retinoids
* Willing to use contraception unless not of childbearing potential
* Able to comply with protocol requirements

Exclusion Criteria:

* Received within 4 weeks prior immunosuppressive medication
* Received treatment within 3 months prior with systemic retinoids (acitretin or isotretinoin)
* Received high potency (class I or II) topical corticoid steroids, topical antibiotics, systemic antibiotics, or topical immunomodulators (tacrolimus or pimecrolimus) within 2 weeks prior to baseline visit
* Received intralesional injections of corticosteroids within 4 weeks prior
* Received surgical intervention for the treatment of HS
* Known history of HIV seropositivity
* History of untreated or active tuberculosis
* Active infection requiring systemic antibiotics within 4 weeks of baseline visit
* History of recurrent/chronic infections
* History of malignancy within 5 years of baseline visit (except for squamous cell carcinoma or basal cell carcinoma; may enroll if treated and assessed as cured).
* Pregnant or breastfeeding
* Immunocompromised due to a medical condition
* Has any significant laboratory abnormalities
* Has any medical condition that may interfere with evaluation of the safety and efficacy of efalizumab
* Received efalizumab or any other biologic within the last 6 months
* Taken or used any investigational drug or device within 30 days prior

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 2005-02; Study Completion 2006-08

PRIMARY OUTCOMES:
Reduction in number of inflammatory lesions 12 weeks post-baseline

SECONDARY OUTCOMES:
Time to the reduction of lesions during 12 weeks of treatment
Percent of disease activity at various weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Strober, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, Dept of Dermatology, New York, New York, United States